CLINICAL TRIAL: NCT01862640
Title: A Phase 3, 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of 2 Fixed Doses of Brexpiprazole (OPC-34712) in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: A Phase 3, 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of 2 Fixed Doses of Brexpiprazole in the Treatment of Alzheimer's Agitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-12-283
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Agitation Associated With; Alzheimer's Disease; Alzheimer's Type; Mental Disorder; Nervous System Diseases
Keywords: OPC-34712; brexpiprazole; Dementia; Alzheimer's Disease; Cognitive Disorders; Agitation
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders; Nervous System Diseases; Dementia; Cognitive Dysfunction; Psychomotor Agitation | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo once daily
  Interventions: Drug: Placebo Oral Tablet
- Brexpiprazole 1 mg (Experimental): Titrate up from 0.25 milligrams (mg)/day brexpiprazole to 1 mg/day brexpiprazole
  Interventions: Drug: Brexpiprazole, OPC-34712
- Brexpiprazole 2 mg (Experimental): Titrate up from 0.25 mg/day brexpiprazole to 2 mg/day brexpiprazole
  Interventions: Drug: Brexpiprazole, OPC-34712

INTERVENTIONS:
Drug: Brexpiprazole, OPC-34712 — Once-daily, tablets
  Arms: Brexpiprazole 1 mg; Brexpiprazole 2 mg
Drug: Placebo Oral Tablet — Once-daily, tablets
  Arms: Placebo

SUMMARY:
To compare the efficacy of 2 fixed doses of brexpiprazole with placebo in participants with agitation associated with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
Behavioral symptoms, such as agitation, are core features in participants with Alzheimer's disease and related dementias and develop in the majority of dementia participants. The presence of agitation in participants with Alzheimer's disease places a significant burden not only on participants and their caregivers but also on the healthcare system.

This is a trial designed to assess the safety and efficacy of brexpiprazole in the treatment of participants with agitation associated with dementia of the Alzheimer's Type. The trial consists of a continuous 12-week double-blind treatment period with a 30-day follow-up. The trial population will include male and female participants between 55 and 90 years of age (inclusive) with a diagnosis of probable Alzheimer's disease, who are residing either in an institutionalized setting or in a non-institutionalized setting where the participant is not living alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 55 to 90 years of age, inclusive, at the time of informed consent.
* Participants who are residing at their current location for at least 14 days before screening and are expected to remain at the same location for the duration of the trial.
* Participants with a diagnosis of probable Alzheimer's disease according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association.
* Participants with a Mini-Mental State Exam score of 5 to 22, inclusive, at screening and baseline visits.
* Participants with onset of symptoms of agitation at least 2 weeks prior to the screening visit.
* Participants with a score of ≥ 4 on the agitation/aggression item of the Neuropsychiatric Inventory-Nursing Home at the screening and baseline visits.
* Participants who require pharmacotherapy for treatment of agitation per the investigator's judgment, after an evaluation for reversible factors (for example, pain, infection, polypharmacy) and a trial of nonpharmacological intervention.
* Participants must have a previous magnetic resonance imaging or computed tomography of the brain, which was performed after the onset of symptoms of dementia, with findings consistent with the diagnosis of Alzheimer's disease.

Exclusion Criteria:

* Participants with dementia or other memory impairment not due to Alzheimer's disease
* Participants with a history of stroke, well-documented transient ischemic attack, pulmonary or cerebral embolism.
* Participants who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, gastrointestinal, or psychiatric disorders.
* Participants who have been diagnosed with an Axis I disorder (Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision criteria)
* Participants with uncontrolled hypertension
* Participants with uncontrolled insulin-dependent diabetes mellitus
* Participants with epilepsy or a history of seizures
* Participants considered in poor general health based on the investigator's judgment.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (66):
- United States (28):
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Bellflower, California
  - Costa Mesa, California
  - Downey, California
  - Orange, California
  - Redlands, California
  - Yorba Linda, California
  - Norwalk, Connecticut
  - Coconut Creek, Florida
  - Hialeah, Florida
  - Lauderhill, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - Sarasota, Florida
  - Decatur, Georgia
  - Suwanee, Georgia
  - Weymouth, Massachusetts
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Mount Arlington, New Jersey
  - Paterson, New Jersey
  - Toms River, New Jersey
  - Hickory, North Carolina
  - Oklahoma City, Oklahoma
  - Franklin, Tennessee
  - Bedford, Texas
  - Waukesha, Wisconsin
- Croatia (3):
  - Rijeka
  - Zadar
  - Zagreb
- Germany (9):
  - Mittweida, Saxony
  - Achim
  - Berlin
  - Bielefeld
  - Bochum
  - Cologne
  - Hamburg
  - Ostfildern
  - Westerstede
- Russia (5):
  - Saint Petersburg
  - Samara
  - Saratov
  - Tonnel’nyy
  - Yekaterinburg
- Serbia (7):
  - Belgrade
  - Kovin
  - Kragujevac
  - Niš
  - Novi Kneževac
  - Novi Sad
  - Vršac
- Spain (8):
  - Barcelona
  - Getafe
  - Girona
  - Madrid
  - Pamplona
  - Salamanca
  - Valencia
  - Zamora
- Ukraine (6):
  - Kharkiv
  - Kherson
  - Kiev
  - Lviv
  - Odesa
  - Poltava

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com

REFERENCES:
- [Derived] Cummings JL, Chumki SR, Chang D, Zhang Z, Brubaker M, Hefting N, Such P, Wang D, Grossberg GT. Efficacy of Brexpiprazole in Participants with Agitation Associated with Dementia Due to Alzheimer's Disease: Pooled Analysis of Randomized Controlled Trials. Clin Drug Investig. 2026 Jan 27. doi: 10.1007/s40261-025-01517-9. Online ahead of print. PMID 41591746
- [Derived] Shah A, Kalu U, Chen D, Slomkowski M, Hobart M, Such P, Grossberg GT. Brexpiprazole side-effect profile in people with agitation in Alzheimer's dementia: a plain language summary. Curr Med Res Opin. 2026 Jan 14:1-3. doi: 10.1080/03007995.2025.2608578. Online ahead of print. PMID 41533472
- [Derived] Grossberg GT, Sabbagh MN, Chumki SR, Wang D, Such P, Zhang Z, Palma AM, Cummings JL. Efficacy of Brexpiprazole on Neuropsychiatric Symptoms and Impact on Caregivers: Pooled Neuropsychiatric Inventory (NPI) Analysis in Patients With Agitation Associated With Dementia due to Alzheimer's Disease. J Geriatr Psychiatry Neurol. 2025 Dec 24:8919887251407124. doi: 10.1177/08919887251407124. Online ahead of print. PMID 41439450
- [Derived] Stroud J, Cummings JL, Chumki SR, Such P, Wang D, Palma AM, Zhang Z, Brubaker M, Grossberg GT. Brexpiprazole for agitation in clinically relevant patient subgroups: a post hoc analysis of efficacy and safety in patients with agitation associated with dementia due to Alzheimer's disease. Curr Med Res Opin. 2025 Aug;41(8):1523-1534. doi: 10.1080/03007995.2025.2552278. Epub 2025 Sep 5. PMID 40847656
- [Derived] Shah A, Estilo A, Sheridan PL, Kalu U, Chen D, Chang D, Slomkowski M, Lee D, Hefting N, Hobart M, Behl S, Such P, Brubaker M, Grossberg GT. Safety and Tolerability of Brexpiprazole in Participants with Agitation Associated with Dementia due to Alzheimer's Disease: Pooled Analysis of Three Randomized Trials and an Extension Trial. CNS Drugs. 2025 Oct;39(10):1011-1023. doi: 10.1007/s40263-025-01200-9. Epub 2025 Jul 19. PMID 40681915
- [Derived] Meunier J, Creel K, Loubert A, Larsen KG, Aggarwal J, Hefting N, Oberdhan D. Defining a clinically meaningful within-patient change threshold for the Cohen-Mansfield Agitation Inventory in Alzheimer's dementia. Front Neurol. 2024 Jul 23;15:1379062. doi: 10.3389/fneur.2024.1379062. eCollection 2024. PMID 39108660
- [Derived] Grossberg GT, Kohegyi E, Mergel V, Josiassen MK, Meulien D, Hobart M, Slomkowski M, Baker RA, McQuade RD, Cummings JL. Efficacy and Safety of Brexpiprazole for the Treatment of Agitation in Alzheimer's Dementia: Two 12-Week, Randomized, Double-Blind, Placebo-Controlled Trials. Am J Geriatr Psychiatry. 2020 Apr;28(4):383-400. doi: 10.1016/j.jagp.2019.09.009. Epub 2019 Oct 1. PMID 31708380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled in this study. The study was conducted in 433 participants at 81 sites in 7 countries: Croatia, Germany, Serbia, Spain, Russia, Ukraine, and the United States.
Pre-assignment Details: Participants attended a screening period ranging from 2 to 42 days. The purpose of the screening period was to determine the participant's eligibility and to washout prohibited concomitant pharmacotherapy prior to randomization.
Groups:
- Brexpiprazole 0.5 mg/Day: All randomized participants received orally brexpiprazole 0.25 milligrams (mg)/day as a starting dose, which was up titrated to 0.5 mg/day. The investigational medicinal product (IMP) was administered once daily in the form of a tablet.
- Brexpiprazole 1 mg/Day: All randomized participants received orally brexpiprazole 0.25 mg/day as a starting dose, which was up titrated to 1 mg/day. The IMP was administered once daily in the form of a tablet.
- Brexpiprazole 2 mg/Day: All randomized participants received orally brexpiprazole 0.25 mg/day as a starting dose, which was up titrated to 2 mg/day. The IMP was administered once daily in the form of a tablet.
- Placebo: All randomized participants received orally brexpiprazole-matching Placebo. The Placebo was administered once daily in the form of a tablet.
Period: Overall Study
Arm/Group | Brexpiprazole 0.5 mg/Day | Brexpiprazole 1 mg/Day | Brexpiprazole 2 mg/Day | Placebo
Started | 20 | 137 | 140 | 136
Completed | 13 | 121 | 122 | 121
Not Completed | 7 | 16 | 18 | 15
Not completed — Adverse Event | 4 | 10 | 6 | 8
Not completed — Participant Met Withdrawal Criteria | 1 | 1 | 2 | 1
Not completed — Participant Withdrawn by Investigator | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 8 | 5
Not completed — Protocol Deviation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 0.5 mg/Day | Brexpiprazole 1 mg/Day | Brexpiprazole 2 mg/Day | Placebo | Total
Number analyzed (Participants) | 20 | 137 | 140 | 136 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (9.1) | 73.8 (8.8) | 73.7 (8.1) | 74.1 (8.0) | 73.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 78 | 79 | 70 | 239
  Male | 8 | 59 | 61 | 66 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 5 | 5 | 12
  White | 20 | 134 | 133 | 130 | 417
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In The Cohen-Mansfield Agitation Inventory (CMAI) Total Score After 12 Weeks Of Brexpiprazole Treatment
Description: To compare the efficacy of 2 fixed doses (1 mg/day and 2 mg/day) of brexpiprazole with placebo in participants with agitation associated with dementia of the Alzheimer's type, by the assessment of CMAI after 12 weeks of treatment. The CMAI assesses the frequency of agitated behaviors in elderly persons, such as hitting, cursing, and restlessness. It consists of 29 items all rated on a 1 to 7 scale with 1 being the "best" rating and 7 being the "worst" rating. The minimum possible CMAI total score is 29, and the maximum possible CMAI total score is 203. A decrease in score indicates improvement in symptoms. To control the overall type I error at 0.05 level when making 2 comparisons of brexpiprazole doses versus placebo, statistical testing was carried out using a hierarchical testing procedure in the order of: 1) comparison of 2 mg/day brexpiprazole versus placebo, and 2) comparison of 1 mg/day brexpiprazole versus placebo.
Time Frame: Baseline, Week 12/Early Termination (ET)
Population: The modified intention-to-treat population consisted of all participants in the randomized sample who took at least 1 dose of IMP (excluding 20 subjects randomized to Brexpiprazole 0.5 mg/day, as doses lower than 1 mg/day were unlikely to be efficacious) and had a baseline and at least 1 post baseline evaluation for the CMAI total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg/Day | Brexpiprazole 1 mg/Day | Placebo
Number analyzed (Participants) | 138 | 134 | 131
units on a scale | -21.6 (1.32) | -17.6 (1.33) | -17.8 (1.34)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day vs Placebo; Test type: Superiority; p = 0.0404, Mixed-effect model repeated measure; Least square (LS) mean difference = -3.77, 95% CI 2-sided [-7.38 to -0.17]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg/Day vs Placebo; Test type: Superiority; p = 0.9015, Mixed-effect model repeated measure; LS mean difference = 0.23, 95% CI 2-sided [-3.40 to 3.86]

2. Secondary Outcome: Change From Baseline In The Clinical Global Impression-Severity Of Illness (CGI-S) Score, As Related To Symptoms Of Agitation After 12 Weeks Of Brexpiprazole Treatment
Description: To compare the efficacy of 2 fixed doses (1 mg/day and 2 mg/day) of brexpiprazole with placebo in participants with agitation associated with Alzheimer's dementia, by the assessment of CGI-S score after 12 weeks of treatment. The CGI-S was used to rate the severity of agitation. Scores were: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. A decrease in score indicates improvement in symptoms.
Time Frame: Baseline, Week 12/ET
Population: The modified intention-to-treat population consisted of all participants in the randomized sample who took at least 1 dose of IMP (excluding 20 participants randomized to Brexpiprazole 0.5 mg/day) and had a baseline and at least 1 post baseline evaluation for the CMAI total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg/Day | Brexpiprazole 1 mg/Day | Placebo
Number analyzed (Participants) | 138 | 134 | 131
units on a scale | -1.29 (1.05) | -1.04 (1.12) | -1.08 (0.89)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day vs Placebo; Test type: Superiority; p = 0.1566, Mixed-effect model repeated measure; LS mean difference = -0.16, 95% CI 2-sided [-0.39 to 0.06]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg/Day vs Placebo; Test type: Superiority; p = 0.4440, Mixed-effect model repeated measure; LS mean difference = 0.09, 95% CI 2-sided [-0.14 to 0.32]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected throughout the study (Baseline to Week 12/ET).
Description: Only participants who received at least 1 dose of study drug were analyzed for safety (Placebo N=135).
Arm/Group | Brexpiprazole 0.5 mg/Day | Brexpiprazole 1 mg/Day | Brexpiprazole 2 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 2/20 | 2/137 | 1/140 | 0/135
Serious Adverse Events (participants affected / at risk) | 5/20 | 11/137 | 13/140 | 7/135
Other Adverse Events (participants affected / at risk) | 11/20 | 27/137 | 43/140 | 29/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 0.5 mg/Day (N=20) | Brexpiprazole 1 mg/Day (N=137) | Brexpiprazole 2 mg/Day (N=140) | Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Intentional Self-Injury (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 0.5 mg/Day (N=20) | Brexpiprazole 1 mg/Day (N=137) | Brexpiprazole 2 mg/Day (N=140) | Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 5 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 2 | 3 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 1 | 1 | 0
Blood Insulin Decreased (Investigations) | 1 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 1 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 1 | 3 | 2 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0 | 0
Protein Total Decreased (Investigations) | 1 | 0 | 0 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 8 | 4
Headache (Nervous system disorders) | 0 | 12 | 13 | 11
Agitation (Psychiatric disorders) | 1 | 2 | 4 | 4
Insomnia (Psychiatric disorders) | 0 | 7 | 8 | 6
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 3
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT01862640/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT01862640/SAP_001.pdf